CLINICAL TRIAL: NCT06390995
Title: A Phase 1/2 Open-label Study to Evaluate The Safety, Tolerability, Efficacy And Pharmacokinetics of Mirvetuximab Soravtansine (TAK-853) in Japanese Patients With Folate Receptor Alpha-Positive Advanced Ovarian Cancer And Other Solid Tumors
Brief Title: A Study of TAK-853 in Adult Participants With Folate Receptor Alpha-Positive Advanced Ovarian Cancer And Other Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-853-1501; jRCT2031240057 (Registry Identifier: jRCT)
Record Dates: First submitted 2024-04-26; First posted 2024-04-30 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Ovarian Cancer; Solid Tumors
MeSH Terms: conditions — Ovarian Neoplasms | interventions — mirvetuximab soravtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phase 1 Part and Phase 2 Part: TAK-853 (Experimental): TAK-853, 6.0 mg/kg, injection, intravenously (IV), once every 3 weeks. Patients will continue to receive study drug until disease progression, unacceptable toxicity, withdrawal of consent, death, or until the sponsor terminates the study (whichever comes first).
  Interventions: Drug: TAK-853

INTERVENTIONS:
Drug: TAK-853 — TAK-853 intravenous injection
  Other Names: Mirvetuximab Soravtansine

SUMMARY:
The main aim of this study are to check for side effects from TAK-853, check how much TAK-853 participants can receive without getting side effects from it, check how well TAK-853 controls symptoms, and to check how much TAK-853 stays in their blood over time.

The study will be conducted in two phases including Phase 1 Part and Phase 2 Part. In Phase 1 Part, the participants will stay in the hospital for 3 days at least after their 1st injection for some tests and to check for any side effects from their treatment. In Phase 2 Part, participants will visit their study hospital for multiple times. In both phases, the participants will receive TAK-853 on the first days of each 3-week cycle.

The participant will be in the study for about 9 months in Phase 1 Part and for about 24 months in Phase 2 Part. The study doctors will check for side effects from the study treatments.

ELIGIBILITY:
Inclusion Criteria:

Phase 1 part:

1. Diagnosis, allowable prior therapy, and disease measurability requirements:

   1. All participants must have a pathologically documented, following advanced solid tumor known to express folate receptor alpha (FR alpha), that is resistant or refractory to standard treatment, for which no standard treatment is available, or the participant refuses standard therapy.

      * Ovarian cancer
      * Endometrial cancer
      * Non-small cell lung cancer (NSCLC)
      * Triple-negative breast cancer (TNBC)
      * Cholangiocarcinoma
      * Colorectal cancer (CRC)
      * Gastro-esophageal adenocarcinoma Note: Participants with a solid tumor type other than the above will be eligible as long as there is prior documentation of tumor FR alpha expression.
   2. All participants without prior documentation of tumor FR alpha expression by immunohistochemistry (IHC) must be willing to provide an archival tumor tissue block or slides, or undergo procedure to obtain a new biopsy using a low risk, medically routine procedure for IHC confirmation of FR alpha positivity of >=1% of viable tumor cells with membrane staining at >=1+ intensity for entry into Phase 1 part
   3. There is no upper limit on the number of prior cytotoxic or targeted therapies the participant may have received. Participants may have received prior treatment with investigational compounds targeting folate receptor excluding MIRV.
   4. Participants must have measurable or non-measurable disease (such as large abdominal masses that cannot be accurately measured) according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
2. Participant must have an Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1
3. Time from Prior Therapy:

   * Systemic anti-neoplastic therapy: five half-lives or four weeks, whichever is shorter (6 weeks for prior nitrosoureas or mitomycin C)
   * FR alpha-targeted therapy: five half-lives or four weeks, whichever is longer
   * Radiotherapy: wide-field radiotherapy (e.g. affecting at least 30% of the bone marrow) completed at least four weeks, or focal radiation completed at least two weeks, prior to starting study drug
4. Participants must have stabilized or recovered (Grade 1 or baseline) from all prior therapy-related toxicities
5. Major surgery must be completed four weeks prior to first dose of TAK-853. Participants must have recovered or stabilized from the side effects prior to study treatment.
6. Participants must have adequate hematologic, liver and kidney function as defined by the following parameters:

   1. Absolute neutrophil count (ANC) >= 1.5*10^9/L (1,500/microliter) without granulocyte colony stimulating factor (G-CSF) in the prior 10 days or long-acting white blood cell (WBC) growth factors in the prior 20 days
   2. Platelet count >= 100.0*10^9/L (100,000/microliter; without platelet transfusion in the prior 10 days)
   3. Hemoglobin >= 9.0 g/dL without packed red blood cell (PRBC) transfusion in the prior 21 days
   4. Serum creatinine =< 1.5* upper limit of normal (ULN) or estimated creatinine clearance of >= 30 mL/minute (as calculated using the Cockcroft Gault equation),
   5. Aspartate aminotransferase (AST) =< 2.5* ULN; alanine aminotransferase (ALT) =< 2.5* ULN (AST, ALT < 5* ULN if liver metastases), and
   6. Total bilirubin =< 1.5* ULN (participants with documented diagnosis of Gilbert syndrome are eligible if total bilirubin < 3.0* ULN)
7. Participants with central nervous system (CNS) disease involvement are eligible if they have had brain metastases resected or have received radiation therapy ending at least 4 weeks prior to study Day 1 and they meet all of the following criteria:

<!-- -->

1. Residual neurological symptoms =< Grade 1
2. No dexamethasone requirement, and
3. Follow-up MRI shows no progression of treated lesions and no new lesions appearing.

Phase 2 part:

1. Participants must have a confirmed diagnosis of high-grade serous epithelial ovarian cancer, primary peritoneal cancer, or fallopian tube cancer
2. Participants must have platinum-resistant disease:

   1. Participants who have only had 1 line of platinum-based therapy must have received at least 4 cycles of platinum, must have had a response (complete response [CR] or partial response [PR]) and then progressed between > 3 months and =< 6 months after the last dose date of platinum
   2. Participants who have received 2 or 3 lines of platinum therapy must have progressed on or within 6 months after the date of the last dose of platinum Note: Progression should be calculated from the date of the last administered dose of platinum therapy to the date of the radiographic imaging showing progression Note: Participants who are primary platinum-refractory during front-line treatment are excluded (see exclusion criteria)
3. Participants must have progressed radiographically on or after their most recent line of therapy
4. Participants must be willing to provide an archival tumor tissue block or slides, or undergo procedure to obtain a new biopsy using a low risk, medically routine procedure for IHC confirmation of FR alpha expression (reported as "positive") as defined by the Ventana FOLR1 Assay. Tumors must be confirmed FR alpha-high as defined by FR alpha positivity of >=75% of viable tumor cells with membrane staining at >=2+ intensity for entry into the Phase 2.
5. Participants must have at least one lesion that meets the definition of measurable disease by RECIST v1.1 criteria (radiologically measured by the Investigator).
6. Participants must have received at least 1 but no more than 3 prior systemic lines of anticancer therapy, and for whom single-agent therapy is appropriate as the next line of treatment:

   a. Neoadjuvant +- adjuvant considered one line of therapy b. Maintenance therapy (e.g., bevacizumab, poly-ADP ribose polymerase [PARP] inhibitors) will be considered as part of the preceding line of therapy (i.e., not counted independently) c. Therapy changed due to toxicity in the absence of progression will be considered as part of the same line (i.e., not counted independently) d. Hormonal therapy will be counted as a separate line of therapy unless it was given as maintenance
7. Participant must have an ECOG PS of 0 or 1
8. Time from prior therapy:

   1. Systemic antineoplastic therapy (5 half-lives or 4 weeks, whichever is shorter)
   2. Focal radiation completed at least 2 weeks prior to first dose of study drug
9. Participants must have stabilized or recovered (Grade 1 or baseline) from all prior therapy-related toxicities
10. Major surgery must be completed at least 4 weeks prior to first dose and the participant must have recovered or stabilized from the side effects of prior surgery
11. Participants must have adequate hematologic, liver, and kidney functions defined as:

    1. ANC >= 1.5* 10^9/L (1,500/microliter) without G-CSF in the prior 10 days or long-acting WBC growth factors in the prior 20 days
    2. Platelet count >= 100* 10^9/L (100,000/microliter) without platelet transfusion in the prior 10 days
    3. Hemoglobin >= 9.0 g/dL without PRBC transfusion in the prior 21 days
    4. Serum creatinine =< 1.5* ULN or estimated creatinine clearance of >= 30 mL/minute (as calculated using the Cockcroft Gault equation).
    5. AST and ALT =< 3.0* ULN
    6. Total bilirubin =< 1.5* ULN (participants with documented diagnosis of Gilbert syndrome are eligible if total bilirubin < 3.0* ULN)
    7. Serum albumin >= 2 g/dL

Exclusion Criteria:

Phase 1 part:

1. Participant with > Grade 1 peripheral neuropathy per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0
2. Participants with active or chronic corneal disorders, history of corneal transplantation, or active ocular conditions requiring ongoing treatment/monitoring such as uncontrolled glaucoma, wet age-related macular degeneration requiring intravitreal injections, active diabetic retinopathy with macular edema, macular degeneration, presence of papilledema, and/or monocular vision.
3. Serious concurrent illness, including, but not limited to the following:

   1. Clinically relevant active infection including - Active hepatitis B or C infection (whether or not on active antiviral therapy)

      - Human Immunodeficiency Virus (HIV) infection

      - Active cytomegalovirus infection

      - Active COVID-19/SARS-CoV-2 infection. Although SARS-CoV-2 testing is not mandatory for study entry, testing should follow local clinical practice guidelines and standards

      - Any other known concurrent infectious disease requiring IV antibiotics within 2 weeks before starting study drug Note: Testing at screening for hepatitis is required, while not required for the remaining infections above unless clinically indicated. Participants with known hepatitis B surface antigen seropositivity and/or detectable hepatitis C virus RNA will be excluded. Participants who have positive hepatitis B core antibody and/or hepatitis B surface antibody can be enrolled but must have an undetectable serum hepatitis B virus DNA. Participants who have positive hepatitis C virus antibody must have an undetectable hepatitis C virus RNA serum level. Participants will be monitored and managed according to Guideline for the prevention of immunosuppressive therapy or chemotherapy-induced reactivation of hepatitis B virus infection (The Japan Society of Hepatology 2022).
   2. Participants with clinically significant cardiac disease including, but not limited to, any one of the following:

      - Myocardial infarction =< 6 months prior to first dose of study medication

      - Unstable angina pectoris

      - Uncontrolled congestive heart failure (New York Heart Association > class II)

      - Uncontrolled >= Grade 3 hypertension (per NCI CTCAE v5.0)

      - Uncontrolled cardiac arrhythmias

      - Severe aortic stenosis
      * >= Grade 3 cardiac toxicity following prior chemotherapy
   3. History of multiple sclerosis or other demyelinating disease, Lambert-Eaton syndrome (paraneoplastic syndrome), history of hemorrhagic or ischemic stroke within the last six months, or alcoholic liver disease.
   4. Previous clinical diagnosis of interstitial lung disease (ILD), including pneumonitis.
4. Any other concomitant anti-cancer treatment such as immunotherapy, biotherapy, radiotherapy, chemotherapy, investigative therapy, or high-dose steroids; however, low-dose steroids and Luteinizing Hormone Releasing Hormone (LHRH) at doses that have been stable for >= 14 days are permitted for participants with prostate cancer
5. Known hypersensitivity to previous monoclonal antibody therapy or maytansinoids, or study drugs and/or any of their excipients
6. Prior history of solid tumor malignancy within the last 3 years except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, in situ breast cancer, in situ prostate cancer (participants must have shown no evidence of active disease for 2 years prior to enrollment)
7. Participants with required use of folate-containing supplements (e.g., folate deficiency)
8. Participants who have received prior allogeneic or autologous bone marrow transplants

Phase 2 part:

1. Participants with endometrioid, clear cell, mucinous, or sarcomatous histology, mixed tumors containing any of the above histologies, or low-grade or borderline ovarian tumor
2. Participants with primary platinum-refractory disease, defined as disease that did not respond to (CR or PR) or has progressed within 3 months of the last dose of first line platinum-containing chemotherapy
3. Participants with prior wide-field radiotherapy affecting at least 20% of the bone marrow
4. Participants with > Grade 1 peripheral neuropathy per NCI CTCAE v5.0
5. Participants with active or chronic corneal disorders, history of corneal transplantation, or active ocular conditions requiring ongoing treatment/monitoring such as uncontrolled glaucoma, wet age-related macular degeneration requiring intravitreal injections, active diabetic retinopathy with macular edema, macular degeneration, presence of papilledema, and/or monocular vision
6. Participants with serious concurrent illness or clinically relevant active infection, including, but not limited to the following:

   1. Active hepatitis B or C infection (whether or not on active antiviral therapy)
   2. HIV infection
   3. Active cytomegalovirus infection
   4. Active COVID-19/SARS-CoV-2 infection. Although SARS-CoV-2 testing is not mandatory for study entry, testing should follow local clinical practice guidelines and standards.
   5. Any other concurrent infectious disease requiring IV antibiotics within 2 weeks before starting study drug Note: Testing at screening for hepatitis (a) is required, while not required for the remaining infections above (b-e) unless clinically indicated.

Participants with known hepatitis B surface antigen seropositivity and/or detectable hepatitis C virus RNA will be excluded. Participants who have positive hepatitis B core antibody and/or hepatitis B surface antibody can be enrolled but must have an undetectable serum hepatitis B virus DNA.

Participants who have positive hepatitis C virus antibody must have an undetectable hepatitis C virus RNA serum level. Participants will be monitored and managed according to Guideline for the prevention of immunosuppressive therapy or chemotherapy-induced reactivation of hepatitis B virus infection (The Japan Society of Hepatology 2022).

7. Participants with history of multiple sclerosis or other demyelinating disease and/or Lambert-Eaton syndrome (paraneoplastic syndrome) 8. Participants with clinically significant cardiac disease including, but not limited to, any one of the following:

1. Myocardial infarction =< 6 months prior to first dose of study medication
2. Unstable angina pectoris
3. Uncontrolled congestive heart failure (New York Heart Association > class II)
4. Uncontrolled >= Grade 3 hypertension (per NCI CTCAE v5.0)
5. Uncontrolled cardiac arrhythmias 9. Participants with a history of hemorrhagic or ischemic stroke within six months prior to first dose of TAK-853 10. Participants with a history of cirrhotic liver disease (Child-Pugh Class B or C) 11. Participants with a previous clinical diagnosis of ILD, including pneumonitis 12. Participants with required use of folate-containing supplements (e.g., folate deficiency) 13. Participants with prior hypersensitivity to monoclonal antibodies or maytansinoids 14. Participants with prior treatment with TAK-853 or other FR alpha-targeting agents 15. Participants with untreated or symptomatic CNS metastases 16. Participants with a history of other malignancy within 3 years prior to first dose of TAK-853 Note: does not include tumors with a negligible risk for metastasis or death (e.g., adequately controlled basal-cell carcinoma or squamous-cell carcinoma of the skin, or carcinoma in situ of the cervix or breast) 17. Prior known hypersensitivity reactions to study drugs and/or any of their excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-04-16 (Actual); Study Completion 2027-03-19 (Estimated)

PRIMARY OUTCOMES:
Phase 1 Part: Number of Participants with Dose-Limiting Toxicities (DLTs) in Cycle 1 | Up to 21 days
  Toxicity will be evaluated according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 5.0. DLT will be defined as any of the events specified in the protocol that are considered by the investigator to be at least possibly related to therapy with study medications.
Phase 1 Part: Number of Participants with Treatment-emergent Adverse Events (TEAEs) | 1 year
  An adverse event (AE) means any untoward medical occurrence in a participant administered a pharmaceutical product; the untoward medical occurrence does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not it is related to the medicinal product. This includes any newly occurring event, or a previous condition that has increased in severity or frequency since the administration of study drug.
Phase 1 Part: Number of Participants with Grade 3 or Higher TEAEs | 1 year
  A severity grade is defined by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0. Grade 1 scales as Mild (asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated); Grade 2 scales as Moderate (minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living [ADL]); Grade 3 scales as Severe (severe or medically significant but not immediately life threatening hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL); Grade 4 scales as Life-threatening consequences, urgent intervention indicated, and Grade 5 scales as Death related to Adverse Event (AE).
Phase 1 Part: Number of Participants with Serious TEAEs | 1 year
  An SAE is any untoward medical occurrence or effect that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability / incapacity, is a congenital anomaly / birth defect or is medically important due to other reasons than the above mentioned criteria.
Phase 1 Part: Number of Participants with TEAEs Leading to Drug Discontinuation. | 1 year
Phase 1 Part: Number of Participants with TEAEs Leading to Infusion Interrupted | 1 year
Phase 1 Part: Number of Participants with TEAEs Leading to Dose Delayed | 1 year
Phase 1 Part: Number of Participants with TEAEs Leading to Dose Reduction | 1 year
Phase 1 Part: Number of Participants with Adverse Event of Clinical Interest (AECIs) | 1 year
  An AE of clinical interest (serious or nonserious) is one of scientific and medical concern specific to the TAK-853, for which ongoing monitoring. Such events may require further investigation to characterize and understand them. AECIs for TAK-853 include: Ocular AEs, Pneumonitis, Peripheral neuropathy, and Infusion related reactions
Phase 2 Part: Overall Response Rate (ORR) Assessed by Investigator with RECIST 1.1 | 2 year
  The ORR is defined as the percentage of participants who achieved a confirmed Partial response (PR) or confirmed Complete response (CR) during the study using RECIST v1.1. Disease response criteria on RECIST 1.1 are following; Complete response (CR): Disappearance of all target lesions. Partial response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. Progressive disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of 1 or more new lesions. Stable disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.

SECONDARY OUTCOMES:
Phase 1 Part: Cmax: Maximum Observed Plasma Concentration | 1 year
  Cmax in Phase 1 Part for intact antibody drug conjugate (ADC), Total Antibody (Ab), DM4 and S-methyl DM4 will be reported.
Phase 1 Part: AUC: Area Under the Plasma Concentration-Time Curve | 1 year
  AUC in Phase 1 Part for intact antibody drug conjugate (ADC), Total Antibody (Ab), DM4 and S-methyl DM4 will be reported.
Phase 1 Part: T1/2: Terminal Half-Life | 1 year
  T1/2 in Phase 1 Part for intact antibody drug conjugate (ADC), Total Antibody (Ab), DM4 and S-methyl DM4 will be reported.
Phase 1 Part: CL: Total Clearance | 1 year
  CL in Phase 1 Part for intact antibody drug conjugate (ADC), Total Antibody (Ab), DM4 and S-methyl DM4 will be reported.
Phase 1 Part: Vss: Volume of Distribution at Steady State | 1 year
  Vss in Phase 1 Part for intact antibody drug conjugate (ADC), Total Antibody (Ab), DM4 and S-methyl DM4 will be reported.
Phase 1 Part: Tmax: Time of First Occurrence of Cmax | 1 year
  Tmax in Phase 1 Part for intact antibody drug conjugate (ADC), Total Antibody (Ab), DM4 and S-methyl DM4 will be reported.
Phase 1 Part: Number of Participants with Immunogenicity of TAK-853 | 1 year
Phase 2 Part: Duration of Response (DOR) Assessed by Investigator with RECIST 1.1 | 2 year
  DOR is defined as the time from the date of the first response (CR or PR), whichever occurs first, to the date of PD or death from any cause, whichever occurs first. DOR Responders without documentation of progressive disease will be censored at the date of last response assessment that is SD or better.
Phase 2 Part: Observed Plasma Concentration | 2 year
  Observed plasma concentration in Phase 2 Part for intact antibody drug conjugate (ADC), Total Antibody (Ab), DM4 and S-methyl DM4 will be reported.
Phase 2 Part: Number of Participants with Immunogenicity of TAK-853 | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (20):
- Japan (20):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - Jikei University Kashiwa Hospital, Kashiwa, Chiba
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Shikoku Cancer Center, Matsuyama, Ehime
  - Kurume University Hospital, Kurume, Fukuoka
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Hyogo Cancer Center, Akashi, Hyōgo
  - Iwate Medical University Hospital, Shiwa-gun, Iwate
  - Tohoku University Hospital, Sendai, Miyagi
  - Saitama Medical University International Medical Center, Hidaka, Saitama
  - Shizuoka Cancer Center, Nakatogari, Shizuoka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Cancer Institute Hospital of JFCR, Koto-ku, Tokyo
  - The Jikei University Hospital, Minato-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Chiba University Hospital, Chiba
  - Kyoto University Hospital, Kyoto
  - Okayama University Hospital, Okayama
  - Osaka International Cancer Institute, Osaka

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/c7b73bd71cf5483b